CLINICAL TRIAL: NCT05225038
Title: Randomized Clinical Trial Investigating Multidimensional Prehabilitation in Pancreatic Surgery for Patients With Pancreatic and Periampullary Neoplasms
Brief Title: Multidimensional Prehabilitation in Pancreatic Surgery for Pancreatic and Periampullary Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8221
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Neoplasms; Periampullary Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Exercise; Behavioral Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Standard of Care) (Active Comparator): Participants will receive the current standard preoperative education and counseling. Participants will receive information regarding exercise and nutrition from a member of the surgical team. Participants will meet with a behavioral medicine specialist for additional education regarding factors affecting postoperative stress and relaxation techniques. Participants who are actively smoking will be counseled regarding smoking cessation and offered a referral to smoking cessation resources.
  Interventions: Behavioral: Behavioral Medicine; Behavioral: Smoking Cessation
- Intervention Arm (Prehabilitation) (Experimental): Participants in the intervention arm will receive all of the standard of care, as listed above, as well as individualized exercise and nutritional prehabilitation regimens.
  During the data analysis, participants will be subdivided into treatment groups, upfront surgical resection versus neoadjuvant chemotherapy, in order to determine whether length of prehabilitation affected outcomes and distinguish any possible effect of chemotherapy toxicity.
  Interventions: Other: Exercise; Dietary Supplement: Nutritional; Behavioral: Behavioral Medicine; Behavioral: Smoking Cessation

INTERVENTIONS:
Other: Exercise — Participants will meet with an exercise physiologist to undergo evaluation and develop individualized regimens for prehabilitation.
  Arms: Intervention Arm (Prehabilitation)
Dietary Supplement: Nutritional — Participants will meet with a nutritionist to undergo evaluation and develop individualized regimens for prehabilitation.
  Arms: Intervention Arm (Prehabilitation)
Behavioral: Behavioral Medicine — Participants will have 1 appointment with behavioral medicine - all participants will meet with the same behavioral medicine specialist to ensure consistency. Participants will receive education regarding factors that affect postoperative recovery and relaxation techniques.
  Participants will also have the option to request faith support.
Behavioral: Smoking Cessation — Participants who are actively smoking will be counseled regarding smoking cessation during their preoperative appointment with a member of the surgical team. They will also be offered a referral to smoking cessation resources.

SUMMARY:
Randomized Clinical Trial Investigating Multidimensional Prehabilitation in Pancreatic Surgery for participants with Pancreatic and Periampullary Neoplasms

DETAILED DESCRIPTION:
Frailty is independently associated with an increased risk of adverse outcomes after major surgery, including pancreatic resection. Prehabilitation aims to optimize modifiable risk factors to improve participants' baseline health prior to surgery. Multiple studies with participants undergoing pancreatic surgery have investigated the impact of prehabilitation on preoperative health metrics as well as postoperative outcomes. The majority of these studies focused only on exercise; if nutritional and/or psychological status were assessed, these dimensions were not intervened upon in prehabilitation regimens or reassessed postoperatively. This randomized controlled trial (RCT) is designed to assess the impact of physical and nutritional prehabilitation on participants' perioperative condition for those undergoing pancreatic resection for diagnosed or suspected pancreatic and periampullary neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Participants > 18 years old with ECOG performance status 0-2 and ASA score ≤3
* Requiring pancreatic resection for diagnosed or suspected pancreatic and periampullary neoplasms
* Surgery scheduled at least 2 weeks after the initial surgical evaluation
* Fluency in English

  * Willingness to answer questionnaires, complete daily exercise & nutrition log, as well as participate in follow-up telephone calls
* Screening: Physical Activity Readiness - Questionnaire (PAR-Q+)

  * PAR-Q+ assesses participants comorbidities and symptoms with current activities. If participants answer "yes" to any of the screening questions, they will need to complete additional questions regarding their chronic medical conditions including, but not limited to, heart disease, stroke, diabetes, depression/anxiety, and COPD/asthma, to determine their ability to participate in physical activity.

Exclusion Criteria:

* Screening: Physical Activity Readiness - Questionnaire (PAR-Q+)

  * Participants with concurrent medical conditions that prohibit exercise, such as those who indicate on the questionnaire that they experience chest pain, dizziness, or loss of consciousness with physical activity; those with chest pain at rest; or those with bone/joint/soft tissue conditions that could worsen with physical activity. Participants with specific comorbidities, such as coronary artery disease. congestive heart failure, or uncontrolled asthma/COPD, that may prevent participation will also be excluded.
* Inability to provide own informed consent
* Inability to read or verbally understand questionnaires in English
* Impaired hearing that creates a barrier for telephone follow-up
* Visual deficit that would cause exercise to be hazardous
* Emergent or urgent surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in participants physical capacity, as represented by hand grip strength | 3 weeks after the surgery
  Previous studies have demonstrated that grip strength is a predictor of surgical outcomes and mortality in cancer participants. Grip strength will be measured utilizing the Jamar Dynamometer.

SECONDARY OUTCOMES:
Mortality Rate | Up to 90 days after the surgery
  Death due to any cause postoperatively.
Morbidity rate | Up to 90 days after the surgery
  Classified according to the Clavien-Dindo Classification of postoperative complications.
Physical capacity as represented by 30s CST (Chair Stand Test ) | 3 weeks after the surgery
  Participants rise to full standing position from sitting in a chair as many times as possible within 30 seconds. The 30s CST has been utilized as a reliable test of lower extremity strength.
Physical capacity as represented by 6-Minute Walk Test | 3 weeks after the surgery
  Participants will walk as far as possible in 6 min at a comfortable pace but do not run or jog. If participants cannot complete the full 6 min walk, then record the time and distance walked and the reason for stopping early.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States